CLINICAL TRIAL: NCT03904446
Title: A Randomized Controlled Trial to Assess the Effectiveness of Multimodal Prophylactic Uterotonics in Patients Undergoing Non-Elective Cesarean Sections After a Trial of Labor
Brief Title: Multimodal Uterotonics at the Time of Cesarean Section in Laboring Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cynthia Wong (Other)
Responsible Party: Sponsor-Investigator, Cynthia Wong, Physician-Professor-DEO, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201904756
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Results first posted 2022-07-27 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Uterine Atony With Hemorrhage
Keywords: Methergine; Uterine Atony
MeSH Terms: conditions — Uterine Inertia | interventions — Methylergonovine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methylergonovine 0.2 mg (Experimental): Standard Oxytocin Infusion at the time of Cesarean Section plus 0.2 mg of Intramuscular Methergine
  Interventions: Drug: Methylergonovine
- Placebo (Normal Saline) (Placebo Comparator): Standard Oxytocin Infusion at the time of Cesarean Section plus 1 milliliter (mL)of normal saline given intramuscular
  Interventions: Drug: Normal Saline (placebo)

INTERVENTIONS:
Drug: Methylergonovine — 0.2 mg of intramuscular methylergonovine at the time of cesarean section following standard IV oxytocin infusion.
  Other Names: Methergine
  Arms: Methylergonovine 0.2 mg
Drug: Normal Saline (placebo) — 1 ml of normal saline intramuscular at the time of cesarean section following standard IV oxytocin infusion
  Other Names: Saline
  Arms: Placebo (Normal Saline)

SUMMARY:
Postpartum hemorrhage remains a leading cause of maternal morbidity and mortality worldwide, even in high income countries. Uterine atony is estimated to cause 70-80% of postpartum hemorrhage. Prolonged labor and augmented labor are known risk factors for postpartum hemorrhage. In attempts to reduce the incidence of postpartum hemorrhage, particularly in patients with known risks factors, it is essential to optimize preventative practices in order to reduce the rates postpartum hemorrhage.

Although oxytocin is considered the first line therapy for preventing and treating uterine atony, early consideration of additional prophylactic uterotonic agents may be indicated in women with prior oxytocin exposure given oxytocin receptor desensitization and down regulation.

As such, investigators sought to examine whether multimodal prophylactic uterotonics (standard oxytocin + methylergonovine), in patients who are increased risk of developing postpartum hemorrhage (specifically laboring patients who ultimately require a cesarean section) would benefit from the addition of prophylactic uterotonics. The clinical rational for administration of multimodal prophylactic uterotonics at the time of cesarean delivery in laboring patients is three-fold: to decrease the incidence of uterine atony, to decrease the incidence of postpartum hemorrhage, decrease the number of uterotonics required at the time of cesarean section.

The primary outcome will be to evaluate the need for additional uterotonic agents (Methylergonovine, Carboprost, Misoprostol) at the time of delivery.

Secondary outcomes will include the incidence of postpartum hemorrhage (quantitative blood loss >1 liter), surgical assessment of uterine tone four minutes following delivery of the placenta, preoperative and postoperative hemoglobin, the need for a blood transfusion, intensive care unit admission, uterine infection (endometritis).

DETAILED DESCRIPTION:
All patients who meet eligibility for the study will be consented during their clinic visit or upon arrival to labor and delivery. If patients elect to participate in the study, enrollment in the study will be noted in their sticky note in EPIC (electronic medical record) which will be ready available to all members of the health care team. If patients during the labor process require a cesarean section, the anesthesiologist will pick up a sealed envelope (which will contain the allocation sequence and group assignment). A randomization block design with mixed block sizes will be used to generate the allocation sequence by using the nQuery Advisor computer software.

The sealed envelopes will be readily available to the anesthesiologist and kept in the anesthesia workroom. Following delivery of the infant, the patient will receive the standard oxytocin infusion. Following administration of the oxytocin infusion, the patient will be given either methylergonovine 0.2 mg IM (intramuscular) or placebo (1 ml of normal saline, intramuscular). This will be drawn up and administered by the anesthesiologist. The obstetrician (delivering provider performing the cesarean section) will be blinded to the group assignment. Documentation of the drug will be recorded in epic in the medication administration record.

The delivering provider will be responsible for determining and relaying to the anesthesiologist whether additional uterotonics are needed throughout the procedure. Additional uterotonics will be given in accordance to the current guidelines outlined by the American Congress of Obstetricians and Gynecologists (ACOG). The delivery provider will assess uterine tone at 4 minutes (satisfactory versus unsatisfactory). The registered nurse will be responsible for setting up a timer to let the OB provider know when 4 minutes have passed. Nursing will call out once the 4 minutes have passed and the OB provider will state whether adequate tone was noted. The anesthesiologist will be responsible for documenting whether a placebo/study drug was given and uterine tone after 4 minutes. This documentation will be placed back into the sealed envelope by the anesthesiologist and placed in the anesthesia workroom. Nicole Masse (primary investigator) will be responsible for storing folders in a secured, locked file cabinet within the Maternal Fetal Medicine offices.

As routinely done at the time of cesarean delivery, the registered nurse will be responsible for measuring and documenting the quantitative blood loss. As routinely performed on all are patients who undergo a vaginal or cesarean delivery, preoperative hemoglobin and postoperative day one hemoglobin levels will be collected.

In the event a postpartum hemorrhage was to occur, the obstetrician will then be un-blinded as management of a postpartum hemorrhage will be driven by whether normal saline or methergine was given as part of the study.

The primary outcome, the need for additional uterotonics, will be assessed in the operating room. Other outcome which will be assessed in the operating room include uterine tone and quantitative blood loss. Outcomes which will be assessed in the immediate postpartum period include: postpartum hemoglobin values, need for a blood transfusion, admission to the intensive care unit, endometritis).

No long-term follow will be needed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Laboring patients who undergo a cesarean section

Exclusion Criteria:

* Placenta/Uterine Abnormalities
* Chronic Hypertension, Gestational Hypertension, Preeclampsia
* HIV/AIDS on protease inhibitors
* History of Coronary Artery Disease
* History of Hypersensitivity to Methylergonovine

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Yes. Pregnant women are the only eligible subjects.
Enrollment: 160 (Actual)
Dates: Start 2019-06-08 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole M Masse, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senturk S, Kagitci M, Balik G, Arslan H, Kir Sahin F. The Effect of the Combined Use of Methylergonovine and Oxytocin during Caesarean Section in the Prevention of Post-partum Haemorrhage. Basic Clin Pharmacol Toxicol. 2016 May;118(5):338-43. doi: 10.1111/bcpt.12500. Epub 2015 Nov 15. PMID 26449959
- [Background] Lavoie A, McCarthy RJ, Wong CA. The ED90 of prophylactic oxytocin infusion after delivery of the placenta during cesarean delivery in laboring compared with nonlaboring women: an up-down sequential allocation dose-response study. Anesth Analg. 2015 Jul;121(1):159-164. doi: 10.1213/ANE.0000000000000781. PMID 25902327
- [Derived] Masse N, Dexter F, Wong CA. Prophylactic Methylergonovine and Oxytocin Compared With Oxytocin Alone in Patients Undergoing Intrapartum Cesarean Birth: A Randomized Controlled Trial. Obstet Gynecol. 2022 Aug 1;140(2):181-186. doi: 10.1097/AOG.0000000000004857. Epub 2022 Jul 6. PMID 35852267

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methylergonovine 0.2 mg | Placebo (Normal Saline)
Started | 80 | 80
Completed | 80 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylergonovine 0.2 mg | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 80 | 160
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 80 | 160
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 80 | 80 | 160

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Need for Additional Uterotonics (Methylergonovine, Carboprost, Misoprostol)
Description: Categorical Variable (Yes/No) - Depending on whether patients required additional uterotonic agents the outcome measure will be yes or no.
Time Frame: Assessed from the time of cesarean section until 24 hours postdelivery
Measure: Count of Participants; unit: Participants
Arm/Group | Methylergonovine 0.2 mg | Placebo (Normal Saline)
Number analyzed (Participants) | 80 | 80
Participants | 80 | 80

2. Secondary Outcome: Quantitative Blood Loss
Description: As per protocol, nurses will measure the quantitative blood loss by measuring the blood in the canisters used during the cesarean section and by weighing the sponges used in the surgery.
Time Frame: Quantitative Blood Loss is measured at the completion of the cesarean delivery, an average of 2 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Methylergonovine 0.2 mg | Placebo (Normal Saline)
Number analyzed (Participants) | 80 | 80
mL | 967 (429) | 1315 (915)

3. Secondary Outcome: The Difference Between the Preoperative and Postoperative (Postpartum Day 1) Hemoglobin Values
Description: As per standard protocol, preoperative and postoperative day one hemoglobin levels will be evaluated. the difference between the preoperative and postoperative day 1 hemoglobin values will be calculated.
Time Frame: Preoperative hemoglobin level is collected on arrival to labor and delivery prior to the cesarean section, postoperative hemoglobin is collected on postoperative day one.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Methylergonovine 0.2 mg | Placebo (Normal Saline)
Number analyzed (Participants) | 80 | 80
g/dL | 2.36 (1.08) | 2.91 (1.08)

4. Secondary Outcome: Number of Patients With Unsatisfactory Uterine Tone 4 Min Following Delivery as Assessed by the Obstetrician
Description: Nursing will notify the obstetrical provider 4 minutes following delivery of the infant and the obstetrical provider will determine whether the uterine tone is noted to be satisfactory (uterus is contracted) or unsatisfactory (uterus boggy)
Time Frame: Obstetricians will assess the uterine tone 4 minutes following delivery of the infant
Measure: Count of Participants; unit: Participants
Arm/Group | Methylergonovine 0.2 mg | Placebo (Normal Saline)
Number analyzed (Participants) | 80 | 80
Participants | 64 | 33

5. Secondary Outcome: The Number of Patients Who Required a Blood Transfusion During the Delivery Hospitalization
Description: The number of patients who required a blood transfusion
Time Frame: The need for a blood transfusion during the cesarean section up until hospital discharge (which is typically postpartum day number 3 for patients undergoing cesarean delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Methylergonovine 0.2 mg | Placebo (Normal Saline)
Number analyzed (Participants) | 80 | 80
Participants | 4 | 18

ADVERSE EVENTS:
Time Frame: During delivery hospitalization (approximately 3-6 days)
Description: Hypertension (defined as blood pressure > 160/110 mmHg)
Arm/Group | Methylergonovine 0.2 mg | Placebo (Normal Saline)
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 7/80 | 9/80
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylergonovine 0.2 mg (N=80) | Placebo (Normal Saline) (N=80)
Hypertension (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 9 (9) — Postpartum diagnosis of pregnancy-induced hypertension

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT03904446/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT03904446/SAP_001.pdf
  • Informed Consent Form (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT03904446/ICF_002.pdf